CLINICAL TRIAL: NCT04351191
Title: Use and Dosage of Hydroxychloroquine and Chloroquine to Convert Symptomatic RT-PCR Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Coronavirus Infectious Disease 2019 (COVID-19) Patients to RT- PCR-Negative as a Means to Reduce Hospitalization Rate
Brief Title: PRophylaxis of Exposed COVID-19 Individuals With Mild Symptoms Using choloroquinE Compounds
Acronym: PRECISE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Government of Punjab, Specialized Healthcare and Medical Education Department (Other Government)
Collaborators: Mayo Hospital Lahore (Other); Services Hospital, Lahore (Other Government); Pakistan Kidney and Liver Institute (Unknown)
Responsible Party: Principal Investigator, Ammar Sarwar, Assistant Professor, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBC-COVID1902
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Sars-CoV2; Symptomatic Condition; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Chloroquine

STUDY DESIGN:
Intervention Model Description: Prospective double blind randomized superiority clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HCQ Regular dose (Active Comparator): Hydroxychloroquine loading dose (400 mg BID for 2 days) followed by 200 mg BID for 4 days plus standard of care
  Interventions: Drug: Hydroxychloroquine Sulfate Regular dose
- HCQ Loading dose (Experimental): Hydroxychloroquine loading dose (400 mg BID) alone plus standard of care
  Interventions: Drug: Hydroxychloroquine Sulfate Loading Dose
- CQ regular dose (Active Comparator): Cholorquine 500 mg BID for 5 days plus standard of care
  Interventions: Drug: Chloroquine
- Placebo (Placebo Comparator): Standard of care plus placebo (cannot be treated with hydroxychloroquine or chloroquine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Regular dose — Hydroxychloroquine administered based off of in-vitro pharmacokinetics study of optimal dosage for efficacy against SARS-CoV-2
  Arms: HCQ Regular dose
Drug: Hydroxychloroquine Sulfate Loading Dose — Hydroxychloroquine administered as a loading dose only
  Arms: HCQ Loading dose
Drug: Chloroquine — Chloroquine administered based off of in-vitro pharmacokinetics study of optimal dosage for efficacy against SARS-CoV-2
  Arms: CQ regular dose
Drug: Placebo — Standard of Care plus placebo
  Arms: Placebo

SUMMARY:
To treat Pakistani patients with non-life threatening symptomatic SARS-CoV-2 infection with an intent to reduce burden on institutional healthcare services by determining efficacy of different chloroquine and hydroxychloroquine dosing regimens in controlling SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patients: defined as fever (temperature greater than 100 degree F), cough, or shortness of breath (respiratory rate >22 per minute).
2. Nasopharyngeal RT-PCR positive SARS-CoV-2
3. Age 20-50 years
4. BMI 18-28 kg/m2
5. Informed consent

Exclusion Criteria:

1. O2 saturation by pulse-oximeter below 93%
2. Co-morbidities: any pre-existing cardiac disease, pulmonary disease, diabetes
3. Arrhythmias and/or history of arrythmia
4. Psoriasis and/or history of psoriasis
5. Neuropathy or myopathy and/or history of these
6. Hypoglycemia and/or history of hypoglycemia
7. Pre-existing hepatic disease
8. Pre-existing renal disease
9. Use of antacids within 1 week
10. Use of antiobiotics within 1 week
11. Pregnancy
12. RT-PCR performed >7 days prior to enrollment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
RT-PCR result | 6th and 7th day
  Percentage of patients who become RT-PCR negative with two RT-PCR tests performed at day 6 and day 7

SECONDARY OUTCOMES:
Progression of symptoms | 7 days
  Time to progression to next stage of SARS-CoV-2 disease severity index
Mortality | 30 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Sarwar, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- Pakistan (4):
  - Expo Covid Isolation Center / Mayo Hospital Field Hospital, Lahore, Punjab Province
  - Mayo Hospital / King Edward Medical University, Lahore, Punjab Province
  - Pakistan Kidney and Liver Institute, Lahore, Punjab Province
  - Services Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No